CLINICAL TRIAL: NCT04891536
Title: Salvage Cryotherapy for Recurrent Prostate Cancer After Brachytherapy or Radiotherapy
Brief Title: Salvage Cryotherapy for Recurrent Prostate Cancer After Radiation Therapy
Acronym: CRIOAND2021
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ignacio Puche Sanz (Other)
Collaborators: Hospital Universitario Reina Sofia de Cordoba (Other Government)
Responsible Party: Sponsor-Investigator, Ignacio Puche Sanz, MD PhD, University Hospital Virgen de las Nieves
Organization: University Hospital Virgen de las Nieves (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRIOAND 0325-N-21
Record Dates: First submitted 2021-05-09; First posted 2021-05-18 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Prostate Cancer; Cryotherapy; Recurrent Prostate Cancer
Keywords: PSMA/PET-CT
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with histologically confirmed recurrent prostate cancer after primary radiation therapy (Experimental)
  Interventions: Procedure: Salvage cryoablation of the prostate (SCAP)

INTERVENTIONS:
Procedure: Salvage cryoablation of the prostate (SCAP) — Cryotherapy of the prostate through transperineal freeezing needles

SUMMARY:
The main objective of this project is to establish a shared comprehensive and systematic protocol for a multicenter prospective registry of patients undergoing salvage cryoablation of the prostate (SCAP).

Our study hypothesis is that SCAP constitutes an effective and safe approach to treat local prostate cancer recurrence after brachytherapy or external beam radiation therapy (EBRT).

DETAILED DESCRIPTION:
Salvage cryoablation of the prostate has been proposed as an alternative to salvage radical prostatectomy, as it has a potentially lower risk of morbidity and equal efficacy. A recent systematic review assessed a total of 32 studies of SCAP (5.513 patients). The overwhelming majority of patients (93%) received whole-gland SCAP. The adjusted pooled analysis for 2-year BCR-free survival for SCAP was 67.49% (95% CI: 61.68-72.81%), and for 5-year BCR-free survival was 50.25% (95% CI: 44.10-56.40%).

Nevertheless, the evidence base relating to the use of SCAP is poor, with significant uncertainties relating to long-term oncological outcomes. One of the main limitations when these studies are analyzed is the lack of information about the histopathology both before starting treatment and at the time of recurrence after cryotherapy. The vast majority only refer to biochemical-free survival as end point, thus limiting interpretation of real oncological performance of this technique. Furthermore, side effects vary widely from study to study and there are uncertainties about the real morbidity associated to cryotherapy in the salvage setting.

Due to this lack of evidence, the EAU 2021 Guidelines recommend that SCAP should only be performed in selected patients in experienced centres as part of a clinical trial or well-designed prospective cohort study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with local recurrence (with histological confirmation) after treatment with radiotherapy or brachytherapy without evidence of distant involvement evaluated with PET/PSMA (if not available then Fluciclovine PET/CT or choline PET/CT must be performed).
* Life expectancy >10 years
* Prostate volume < 100cc
* PSA<10 ng/mL
* mpMRI + fusion/systematic biopsy ≤cT3a without affecting the bladder neck or the membranous urethra

Exclusion Criteria:

* Patients with clinically confirmed distant metastasis
* Any previous major rectal surgery
* Clinically significant lower urinary tract or rectal anomalies
* Existing urethral, rectal, or bladder fistulae

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Disease-free rate | 1 year
  absence of disease in follow-up biopsy AND PET/PSMA
ADT-free survival | 5 years
  Absence of androgen deprivation therapy need during follow-up

SECONDARY OUTCOMES:
Rate of incontinence | 1 year
  Measured by International Consultation on Incontienence Questionnaire short-form (ICIQ-SF)
Rate of sexual disfunction | 1 year
  Measured by International Index Erectile Function (IIEF-25)
Effect on urinary symptoms | 1 year
  Measured by International Prostate Symptoms Score (IPSS) and uroflowmetry
Biochemical free survival | 5 years
  PSA
Metastasis free survival | 5 years
  Metastasis detected in novel imaging modalities
Performance of mpMRI and PET-CT for the detection of clinically significant recurrence. | 1 year
  Related to the histopathology observed
Rate of metastasis detected by PET-CT | 1 year
  Metastais detected

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Hospital Universitario Reina Sofía, Córdoba, Andalusia
  - Hospital Universitario Virgen de las Nieves, Granada, Andalusia

IPD SHARING:
Plan to Share IPD: No